CLINICAL TRIAL: NCT07332962
Title: An Exploratory Clinical Study on fMRI-Based Evaluation of Intervention Targets for Auricular Acupuncture Therapy
Brief Title: fMRI Evaluation of Auricular Acupuncture Targets: An Exploratory Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Principal Investigator, Ming Chu, The deputy dean of the hospital, Jiangsu Taizhou People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: LSKY 2025-175-01
Record Dates: First submitted 2025-12-13; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: fMRI; clinical trial; functional connectivity; auricular press needles
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group used disposable sterile auricular press needles (Experimental)
  Interventions: Device: Effect of Verum Auricular Acupuncture on Resting-State Brain Function in Healthy Subjects: A Functional Magnetic Resonance Imaging (fMRI) Study
- The control group received a needle-free, disposable, sterile auricular press needles. (Sham Comparator)
  Interventions: Device: Sham Auricular Acupuncture as a Control Intervention for Brain fMRI Studies in Healthy Volunteers

INTERVENTIONS:
Device: Effect of Verum Auricular Acupuncture on Resting-State Brain Function in Healthy Subjects: A Functional Magnetic Resonance Imaging (fMRI) Study — The auricular points Heart, Kidney, Shenmen, and Subcortex were selected. After a baseline fMRI scan, sterile press needles were applied aseptically to these points in the experimental group.Each point was stimulated with 20 manual presses per session. This procedure was repeated for three sessions, separated by 10-minute intervals, resulting in a total intervention time of approximately 26 minutes. To capture immediate neural effects, a post-intervention fMRI scan was conducted to observe changes in brain activity.
  The intervention involved applying auricular press needles (a type of intradermal embedding needle) to specific acupoints.
  Arms: The experimental group used disposable sterile auricular press needles
Device: Sham Auricular Acupuncture as a Control Intervention for Brain fMRI Studies in Healthy Volunteers — The sham auricular acupuncture control group was identical to the experimental group in terms of acupoint locations, auricular acupuncture procedure, and fMRI scanning protocol. The sole exception was that the sham group received a needle-free, auricular press needles.
  Arms: The control group received a needle-free, disposable, sterile auricular press needles.

SUMMARY:
This study employs resting-state functional magnetic resonance imaging (rs-fMRI) to examine whether auricular press needles acupuncture modulates functional connectivity between the insula and medial prefrontal cortex (MPFC), in a manner comparable to transcranial vagus nerve stimulation (taVNS), and to assess its association with interoceptive improvement. By establishing a neurophysiological baseline for auricular vagus nerve stimulation (aVNS) in the healthy brain, the research aims to clarify its regulatory mechanisms in cognition and emotion. The findings provide a key theoretical and evaluative framework for translating aVNS into clinical applications for insomnia and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-30 years;
2. Basically normal diet and sleep;
3. No history of mental illness;
4. No MRI contraindications (e.g., metal implants or pacemakers) or claustrophobia；
5. Willing to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Presence of auricular skin lesions or allergy to adhesive ear patches;
2. Currently receiving regular acupuncture treatment;
3. History of bleeding disorders or anticoagulant use (increased bleeding risk);
4. Previous history of syncope during acupuncture.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity strength between the insula and the medial prefrontal cortex (MPFC)(T1-T0) | From enrollment to the end of treatment at 2 weeks
  Data collection is divided into two stages:
  Baseline : Collection of demographic data, baseline fMRI scan, and clinical assessment(T0).
  post-intervention : fMRI scan and clinical assessment immediately after the intervention(T1).
  The functional connectivity between the bilateral insula and medial prefrontal cortex was quantified by calculating the Pearson correlation of their mean time series at baseline and post-intervention. This connectivity strength serves as a proxy for the efficiency of information exchange between the interoceptive hub and the self-referential/emotion-regulatory hub. An increase following auricular acupuncture may reflect enhanced psychosomatic integration and top-down emotional regulation, suggesting a functional optimization of this circuit. Conversely, a decrease could indicate a disruption of pathological hyper-connectivity related to emotional constraint or an upregulation of control-mechanisms consistent with the observed alleviation of emotional symptoms

SECONDARY OUTCOMES:
Local brain activity indicators:regional homogeneity (ReHo)（T1-T0） | From enrollment to the end of treatment at 2 weeks
  Regional homogeneity (ReHo) was calculated as Kendall's coefficient of concordance between each voxel and its 26 nearest neighbors, assessed separately before and after the intervention. This metric captures the temporal synchrony of neural activity within local brain regions. Following auricular acupuncture, increased ReHo in regions such as the insula and prefrontal cortex may reflect improved neural coordination and functional integration. Conversely, decreased ReHo in specific areas could indicate a modulatory effect on abnormally elevated local synchrony.
Local brain activity indicators:amplitude of low-frequency fluctuation (ALFF)（T1-T0） | From enrollment to the end of treatment at 2 weeks
  Amplitude of low-frequency fluctuation (ALFF) was quantified by calculating the square root of the power spectrum within the 0.01-0.08 Hz frequency band of the BOLD signal, followed by normalization to the global mean ALFF value. This metric reflects the intensity of spontaneous neural activity in the brain. An increase in ALFF within emotion- and cognition-related regions following auricular acupuncture may indicate an elevation in baseline neural activity or metabolic activity in these areas. Conversely, a decrease in ALFF in regions such as the limbic system could reflect an inhibitory modulatory effect of the intervention on hyperactivity, potentially contributing to emotional stabilization.
Local brain activity indicators:fractional amplitude of low-frequency fluctuation (fALFF)（T1-T0） | From enrollment to the end of treatment at 2 weeks
  Fractional amplitude of low-frequency fluctuation (fALFF) was quantified by calculating the ratio of low-frequency ALFF to the full-frequency ALFF before and after the intervention, followed by normalization to the global mean fALFF value. Changes in fALFF following the intervention allow a more specific assessment of auricular acupuncture's regulatory effects on intrinsic neural oscillations related to cognition and emotion. When interpreted in conjunction with ALFF changes, the direction of fALFF alteration can help elucidate the specific mechanisms through which auricular acupuncture modulates neural activity patterns.
Interhemispheric coordination index: voxel-mirrored homotopic connectivity (VMHC)（T0-T1） | From enrollment to the end of treatment at 2 weeks
  Voxel-Mirrored Homotopic Connectivity (VMHC) was assessed by calculating the Pearson correlation coefficient between BOLD time series from symmetrically corresponding voxel pairs in the left and right hemispheres, separately before and after the intervention. The VMHC value quantifies the functional coordination between homotopic regions across the two cerebral hemispheres. Following auricular acupuncture, enhanced VMHC in regions associated with emotional regulation and cognitive control, such as the prefrontal cortex and anterior cingulate cortex, may suggest improved interhemispheric balance and integration of emotional processing. Conversely, changes in VMHC within specific regions could help clarify how the intervention modulates functional imbalances between hemispheres, particularly those related to constrained emotional states.

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou People's Hospital affiliated to Nanjing Medical University, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly due to participant privacy/confidentiality restrictions and the terms of the informed consent obtained for this study. Summary data are available upon reasonable request.

REFERENCES:
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Qi M, Huang Y, Mai R, Yan Z, Xu B, Liu B, Zhang Y. Baseline functional connectivity of the basal forebrain-cortical circuit predict taVNS treatment response in primary insomnia: a randomized controlled trial and fMRI study. BMC Med. 2025 Jul 9;23(1):412. doi: 10.1186/s12916-025-04126-7. PMID 40629377
- [Background] Huang Y, Zhang Y, Hodges S, Li H, Yan Z, Liu X, Hou X, Chen W, Chai-Zhang T, Kong J, Liu B. The modulation effects of repeated transcutaneous auricular vagus nerve stimulation on the functional connectivity of key brainstem regions along the vagus nerve pathway in migraine patients. Front Mol Neurosci. 2023 Jun 2;16:1160006. doi: 10.3389/fnmol.2023.1160006. eCollection 2023. PMID 37333617
- [Background] Zhang S, He JK, Meng H, Zhao B, Zhao YN, Wang Y, Li SY, Wang L, Wu MZ, Chen Y, Xiao X, Hou LW, Fang JL, Rong PJ. Effects of transcutaneous auricular vagus nerve stimulation on brain functional connectivity of medial prefrontal cortex in patients with primary insomnia. Anat Rec (Hoboken). 2021 Nov;304(11):2426-2435. doi: 10.1002/ar.24785. Epub 2021 Oct 8. PMID 34623769
- [Background] Ferreira LA, Grossmann E, Januzzi E, Goncalves RT, Mares FA, de Paula MV, Carvalho AC. Ear Acupuncture Therapy for Masticatory Myofascial and Temporomandibular Pain: A Controlled Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:342507. doi: 10.1155/2015/342507. Epub 2015 Aug 17. PMID 26351510
- [Background] Moss DA, Crawford P. Ear Acupuncture for Acute Sore Throat: A Randomized Controlled Trial. J Am Board Fam Med. 2015 Nov-Dec;28(6):697-705. doi: 10.3122/jabfm.2015.06.150014. PMID 26546644
- [Background] Wu S, Liang J, Zhu X, Liu X, Miao D. Comparing the treatment effectiveness of body acupuncture and auricular acupuncture in preoperative anxiety treatment. J Res Med Sci. 2011 Jan;16(1):39-42. PMID 21448381
- [Background] Uddin N, Levine DL. Battlefield Acupuncture for the Treatment of Chronic Migraines. Cureus. 2024 May 15;16(5):e60369. doi: 10.7759/cureus.60369. eCollection 2024 May. PMID 38883138
- [Background] Natbony LR, Zhang N. Acupuncture for Migraine: a Review of the Data and Clinical Insights. Curr Pain Headache Rep. 2020 May 29;24(7):32. doi: 10.1007/s11916-020-00864-w. PMID 32472196
- [Background] de Oliveira Rodrigues DM, Menezes PR, Machado Ribeiro Silotto AE, Heps A, Pereira Sanches NM, Schveitzer MC, Faisal-Cury A. Efficacy and Safety of Auricular Acupuncture for Depression: A Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2345138. doi: 10.1001/jamanetworkopen.2023.45138. PMID 38032640
- [Background] Zhang Y, Lin P, Wang R, Zhou J, Xu X, Jiang W, Pu X, Ge S. Insula-Medial Prefrontal Cortex Functional Connectivity Modulated by Transcutaneous Auricular Vagus Nerve Stimulation: An fMRI Study. IEEE J Biomed Health Inform. 2024 Oct;28(10):5962-5970. doi: 10.1109/JBHI.2024.3423019. Epub 2024 Oct 3. PMID 38963749
- See also: Related Info — https://pubmed-ncbi-nlm-nih-gov-s.atrust.seu.edu.cn/38963749/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT07332962/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT07332962/ICF_001.pdf